CLINICAL TRIAL: NCT05067439
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE, 2-PERIOD STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSE ABROCITINIB ON THE PHARMACOKINETICS OF SINGLE DOSES OF CAFFEINE, EFAVIRENZ, AND OMEPRAZOLE IN HEALTHY PARTICIPANTS
Brief Title: A Study to Estimate the Effect of Multiple Dose Abrocitinib on Caffeine, Efavirenz, and Omeprazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B7451092
Expanded Access: NCT05466578 (Available)
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: abrocitinib; drug-drug interaction; omeprazole; caffeine; efavirenz
MeSH Terms: interventions — abrocitinib; Omeprazole; Caffeine; efavirenz

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 (Other): In Period 1, all the participants will receive single doses of the probe drugs, including caffeine 100 mg, efavirenz 50 mg and omeprazole 10 mg, together on Day 1.
  Interventions: Drug: Omeprazole; Drug: Caffeine; Drug: Efavirenz
- Period 2 (Other): In Period 2, participants will receive abrocitinib 200 mg once daily (QD) on Day 1-10, single dose of omeprazole on Day 2 and single dose of probe drugs together on Day 8.
  Interventions: Drug: Abrocitinib; Drug: Omeprazole; Drug: Caffeine; Drug: Efavirenz

INTERVENTIONS:
Drug: Abrocitinib — 200 mg once daily (QD)
  Arms: Period 2
Drug: Omeprazole — single doses of 10 mg
Drug: Caffeine — single dose of 100 mg
Drug: Efavirenz — single doses of 50 mg

SUMMARY:
This is a Phase 1, open-label, multiple dose, single fixed-sequence, 2-period study to evaluate the effect of abrocitinib on the pharmacokinetics (PK) of caffeine, efavirenz and omeprazole in healthy adult participants. A total of approximately 13 healthy male and/or female participants will be enrolled in the study to obtain at least 12 evaluable participants who complete the study. Participants who withdraw from the study or are considered non-evaluable may be replaced at the discretion of the sponsor. Participants will be screened within 28 days of the first dose of study intervention. Participants will have a phone contact 3 days prior to Day 1 dosing (Day -3) in Period 1 as a reminder to abstain from caffeine-containing products. Participants will be admitted to the clinical research unit (CRU) at least 24 hours prior to Day 1 dosing (Day 1) in Period 1. Participants will remain in the CRU for a total of 15 days and 14 nights. Participants will have a telephone contact between 28-35 calendar days after the last administration of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥18 years of age at the time of signing the Informed consent document (ICD).
2. Male and female participants who are healthy as determined by medical evaluation including a detailed medical history, complete physical examination, laboratory tests, and cardiovascular tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Body mass index (BMI) of 17.5 to 32 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, neurological diseases, or other systems diseases, allergic diseases including drug allergies but excluding untreated asymptomatic seasonal allergies at the time of dosing
2. Subjects with moderate to severe gastroesophageal reflux disease (GERD) symptoms, or any condition affecting drug absorption e.g. gastrectomy, cholecystectomy
3. History of human immunodeficiency virus (HIV) infection, positive test for HIV, hepatitis B, hepatitis C, positive test for hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb). Subjects previously vaccinated for hepatitis B may be allowed. However, subjects vaccinated with vaccines having live or attenuated components within 6 weeks of the first dose of study drug, or expecting to be vaccinated during the course of the trial are excluded.
4. Any psychiatric condition including recent or active suicidal ideation or behavior, other psychiatric conditions that may increase the risk of study participation, or, in the investigator's judgement, make the subject inappropriate for the study.
5. Evidence or history of clinically significant dermatological conditions, e.g. atopic dermatitis (AD) or psoriasis, or visible rash present during physical examination, history of disseminated herpes zoster or disseminated herpes simplex, or localized dermatomal herpes zoster.
6. History of chronic infections, recurrent infections or latent infections, e.g. tuberculosis (TB); Positive QuantiFERONE® TB GOLD test, any acute infection within 2-weeks of baseline (Day-1).
7. Malignancies or history of malignancies except for adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
8. History of hypersensitivity, intolerance, or allergic reaction associated with prior exposure to caffeine, omeprazole, efavirenz and abrocitinib or any of their excipients.
9. Subjects who may be at increased risk if dosed with efavirenz, including severe hepatic impairment (Child Pugh Class C), or a history of seizures.
10. Use of prescription or non-prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study drug; herbal supplements and hormonal contraceptives and hormone replacement therapy (HRT) must be discontinued at least 28 days prior to the first dose of the investigational product; Depo-Provera® must be discontinued at least 6 months prior to dosing with investigational product.
11. Systemic therapy with any of the medicines that are moderate or strong cytochrome P450 (CYP)1A2, CYP2B6, or CYP2C19 inhibitors within 28 days or 5 half-lives (whichever is longer), or moderate or strong CYP1A2, CYP2B6 or CYP2C19 inducers within 28 days or 5-half-lives (whichever is longer) prior to the first dose.
12. Previous administration with any investigational drug within 30 days (or as determined by local requirements), or 5-half-lives preceding the first dose of study drug intervention used in this study (whichever is longer).
13. Smokers and/or subjects who used nicotine-based products within three months prior to the first dose of the investigational product.
14. Screening supine blood pressure (BP)≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at last 5 minutes of supine rest. If BP≥140 mmHg (systolic) or ≥90 mmHg (diastolic), the BP should be repeated 2 more times and the average of the 3BP values should be used to determine the subject's eligibility.
15. Abnormal baseline standard 12-lead electrocardiogram (ECG), QT interval >450 msec, QTcF>450 msec, . If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the subjects eligibility. Computer-interpreted ECGs should be 0ver-read by a physician experienced in reading ECGs before excluding a subject.
16. Subjects with abnormal blood chemistry; abnormal hematology including complete WBC count and differentials; estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 m2
17. History of alcohol abuse, binge drinking, or any illicit drug use or dependence within 6 months of screening. Positive urine drug test.
18. Pregnant females, breastfeeding females, female subjects of childbearing potential who are unwilling or unable to use one highly effective method of contraception as outlined in the protocol for the duration of the study and for at least, 28 days after the last dose of study intervention. Unwilling to comply with lifestyle considerations in the protocol.
19. Subjects who routinely consume more than five 8-ounce cups of coffee (or caffeine equivalent), or greater than 6 servings (1 serving is approximately equivalent to 125 mg of caffeine) of tea, cola or other caffeinated beverage per day.
20. Consumption of chocolate and chocolate-containing products (e.g. hot chocolate, ice cream, cookies, etc) within 48 hours prior to the first dose of study drug and during the study.
21. Consumption of charcoal-broiled beef within 7 days prior to the first dose of study drug as it is known to induce CYP1A2 enzyme.
22. Consumption of cruciferous vegetables (e.g. cauliflower, broccoli, Brussel sprouts and cabbage) within 7 days prior to the first dose of study drug as cruciferous vegetables are known to increase CYP1A2 activity
23. Blood donation (excluding plasma donation) of approximately 1 pint (500 ml) or more within 60 days prior to dosing.
24. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator and their respective family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Research Centers of America ( Hollywood ), Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang X, Dowty ME, Tripathy S, Le VH, Huh Y, Curto M, Winton JA, O'Gorman MT, Chan G, Malhotra BK. Assessment of the Effects of Abrocitinib on the Pharmacokinetics of Probe Substrates of Cytochrome P450 1A2, 2B6 and 2C19 Enzymes and Hormonal Oral Contraceptives in Healthy Individuals. Eur J Drug Metab Pharmacokinet. 2024 May;49(3):367-381. doi: 10.1007/s13318-024-00893-5. Epub 2024 Mar 30. PMID 38554232
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451092

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 26 participants were assigned and dosed in this study. In addition to the initial 13 participants planned, this study enrolled 13 replacement participants due to pharmacokinetic (PK) sample lost and remaining samples being not evaluable. Thus only 13 participants were included in the PK analysis.
Groups:
- Periods 1 and 2: Healthy participants received single oral doses of caffeine 100 mg, efavirenz 50 mg, and omeprazole 10 mg together following an overnight fast on Day 1 Period 1. They received abrocitinib 200 mg orally once daily (QD) on Days 1 - 10 Period 2, a single oral dose of omeprazole 10 mg on Day 2 Period 2, and single oral doses of caffeine 100 mg, efavirenz 50 mg, and omeprazole 10 mg together on Day 8 Period 2.
Period: Period 1
Arm/Group | Periods 1 and 2
Started | 26
Completed | 26
Not Completed | 0
Period: Period 2
Arm/Group | Periods 1 and 2
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study intervention.
Groups:
- Periods 1 and 2: Healthy participants received single oral doses of caffeine 100 mg, efavirenz 50 mg, and omeprazole 10 mg together following an overnight fast on Day 1 Period 1. They received abrocitinib 200 mg orally QD on Days 1 - 10 Period 2, a single oral dose of omeprazole 10 mg on Day 2 Period 2, and single oral doses of caffeine 100 mg, efavirenz 50 mg, and omeprazole 10 mg together on Day 8 Period 2.
Arm/Group | Periods 1 and 2
Number analyzed (Participants) | 26
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0
  18-44 | 16
  45-64 | 10
  >=65 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23
  Black or African American | 3
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26.72 [20.6 to 30.2]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Omeprazole
Description: AUCinf was defined as area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72 hour post-dose on Day 1 Period 1 and Day 8 Period 2
Population: This study enrolled 13 replacement participants as some of the pharmacokinetic (PK) samples from Day 8 Period 2 collected from the initial 13 participants were lost in transit and remaining samples were not evaluable. The PK data collected from the 13 replacement participants were included in the following descriptive and statistical summaries.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg: Healthy participants received single oral doses of caffeine 100 mg, efavirenz 50 mg, and omeprazole 10 mg together following an overnight fast on Day 1 Period 1.
- Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg: Healthy participants received abrocitinib 200 mg orally QD on Days 1 - 10 Period 2 and single oral doses of caffeine 100 mg, efavirenz 50 mg, and omeprazole 10 mg together on Day 8 Period 2.
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
Number analyzed (Participants) | 13 | 13
ng*hr/mL | 238.5 (101) | 688.8 (90)
Statistical Analysis 1: Comparison: Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg vs Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg; Omeprazole 10 mg was Reference and abrocitinib 200 mg + omeprazole 10 mg was Test. Natural log-transformed AUCinf was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect and estimates of the adjusted mean differences (Test-Reference) and 90% CIs were obtained. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI; Test type: Other; Ratio of Adjusted Geometric Means = 288.81, 90% CI 2-sided [240.56 to 346.73]

2. Primary Outcome: AUCinf Corrected for Residual Concentrations (AUCinfCR) of Caffeine
Description: AUCinfCR was defined as AUCinf corrected for residual concentrations. AUCinf was defined as area under the plasma concentration-time profile from time 0 extrapolated to infinite time. Two participants in Period 1 and 1 participant in Period 2 had pre-dose caffeine concentrations that were greater than 5% of the corresponding maximum plasma concentration (Cmax). Therefore, AUCinf was corrected for the residual concentrations for these participants.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72 hour post-dose on Day 1 Period 1 and Day 8 Period 2
Population: This study enrolled 13 replacement participants as some of the PK samples from Day 8 Period 2 collected from the initial 13 participants were lost in transit and remaining samples were not evaluable. The PK data collected from the 13 replacement participants were included in the following descriptive and statistical summaries.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
Number analyzed (Participants) | 12 | 11
ng*hr/mL | 19730 (46) | 26880 (28)
Statistical Analysis 1: Comparison: Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg vs Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg; Caffeine 100 mg was Reference and abrocitinib 200 mg + caffeine 100 mg was Test. Natural log-transformed AUCinfCR was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect and estimates of the adjusted mean differences (Test-Reference) and 90% CIs were obtained. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI; Test type: Other; Ratio of Adjusted Geometric Means = 139.59, 90% CI 2-sided [121.98 to 159.74]

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration Corrected for Residual Concentrations (AUClastCR) of Efavirenz
Description: AUClastCR was defined as AUClast corrected for residual concentrations. AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. Eight participants in Period 2 had pre-dose efavirenz concentrations that were greater than 5% of the corresponding Cmax. Therefore, AUClast was corrected for the residual concentrations for these participants.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72 hour post-dose on Day 1 Period 1 and Day 8 Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
Number analyzed (Participants) | 13 | 13
ng*hr/mL | 5588 (20) | 6153 (24)
Statistical Analysis 1: Comparison: Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg vs Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg; Efavirenz 50 mg was Reference and abrocitinib 200 mg + efavirenz 50 mg was Test. Natural log-transformed AUClastCR was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect and estimates of the adjusted mean differences (Test-Reference) and 90% CIs were obtained. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI; Test type: Other; Ratio of Adjusted Geometric Means = 110.10, 90% CI 2-sided [103.45 to 117.17]

4. Secondary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or worsened relative to pretreatment state. An SAE was defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect.
Time Frame: Up to 48 days after the first dose in period 1. This includes 3 days of period 1, 10 days of period 2 and 28-25 days of the follow-up period.
Population: All 26 participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Abrocitinib 200 mg QD + Omeprazole 10 mg: Healthy participants received abrocitinib 200 mg orally QD on Days 1 - 10 Period 2 and a single oral dose of omeprazole 10 mg on Day 2 Period 2.
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
Number analyzed (Participants) | 26 | 26 | 26
Participants
  TEAEs | 3 | 1 | 5
  SAEs | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-Related TEAEs and SAEs
Description: Adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or worsened relative to pretreatment state. An SAE was defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect. Causality of the TEAEs and SAEs was judged by the investigator.
Time Frame: as for outcome 4
Population: All 26 participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
Number analyzed (Participants) | 26 | 26 | 26
Participants
  TEAEs | 2 | 0 | 1
  SAEs | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities Regardless of Baseline
Description: Hematology parameters included hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet and white blood cell count, total neutrophils, eosinophils, monocytes, basophils and lymphocytes. Chemistry parameters included blood urea nitrogen, cystatin C, glucose (fasting), calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein. Urine parameters included pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy. Only those categories in which at least 1 participant had data were reported. Number of Participants With Laboratory Abnormalities Regardless of Baseline in data table indicates the number of participants who had the laboratory abnormality at least 1 of the timepoints when the laboratory tests were done.
Time Frame: At screening, on Day -1 Period 1 and Day 11 Period 2
Population: All 26 participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
Number analyzed (Participants) | 26 | 26 | 26
Participants
  Neutrophils >1.2x upper limit of normal (ULN) | 0 | 0 | 1
  Urine hemoglobin >=1 | 0 | 0 | 7

7. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs
Description: Vital sign measurements included supine blood pressure, pulse rate, respiratory rate, and temperature. Any safety assessments (vital sign measurements) including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator were considered meeting the AE definition and are listed below. Only those categories in which at least 1 participant had data were reported.
Time Frame: At screening, on Day 1 Period 1 and Day 11 Period 2
Population: All 26 participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
Number analyzed (Participants) | 26 | 26 | 26
Participants | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 48 days after the first dose in period 1. This includes 3 days of period 1, 10 days of period 2 and 28-25 days of the follow-up period.
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Groups:
- Abrocitinib 200 mg QD + Omeprazole 10 mg: Healthy participants received abrocitinib 200 mg orally QD on Days 1 - 10 Period 2, and a single oral dose of omeprazole 10 mg within approximately 5 minutes after administration of abrocitinib on Day 2 Period 2.
Arm/Group | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg | Abrocitinib 200 mg QD + Omeprazole 10 mg | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 2/26 | 0/26 | 3/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg (N=26) | Abrocitinib 200 mg QD + Omeprazole 10 mg (N=26) | Abrocitinib 200 mg QD + Caffeine 100 mg + Efavirenz 50 mg + Omeprazole 10 mg (N=26)
Blood pressure increased (Investigations) | 0 | 0 | 2
Tremor (Nervous system disorders) | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
In addition to the initial 13 participants, this study enrolled 13 replacement participants as some of the PK samples from Day 8 Period 2 collected from the initial 13 participants were lost in transit and remaining samples were not evaluable. This replacement is consistent with the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT05067439/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT05067439/SAP_001.pdf